CLINICAL TRIAL: NCT01141660
Title: Use of Laryngeal Mask Airway in Pediatric Adenotonsillectomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Virginia Commonwealth University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HM10692
Record Dates: First submitted 2010-06-07; First posted 2010-06-10 (Estimated); Results first posted 2011-01-13 (Estimated); Last update posted 2017-11-13 (Actual); Status verified 2017-10

CONDITIONS: Laryngeal Mask Airway; Tonsillectomy
MeSH Terms: interventions — Intubation, Intratracheal; Laryngeal Masks

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Endotracheal Tube (Experimental): Children undergoing adenotonsillectomy are randomized to endotracheal tube or laryngeal mask airway.
  Interventions: Device: Endotracheal Tube
- Laryngeal Mask Airway (Experimental): Children undergoing adenotonsillectomy are randomized to endotracheal tube or laryngeal mask airway.
  Interventions: Device: Laryngeal mask airway

INTERVENTIONS:
Device: Endotracheal Tube — Patients randomized to either Laryngeal Mask Airway or Endotracheal tube prior to undergoing adenotonsillectomy.
  Other Names: ETT; Endotracheal intubation
  Arms: Endotracheal Tube
Device: Laryngeal mask airway — Randomized to either Laryngeal mask airway or endotracheal tube
  Other Names: LMA
  Arms: Laryngeal Mask Airway

SUMMARY:
The aim of the current study is to compare the use of laryngeal mask airway (LMA) and endotracheal tube (ETT) in pediatric adenotonsillectomy. The primary objective is to assess the incidence of post-operative laryngospasm between the LMA and ETT. The investigators also sought to compare anesthetic, operative, and recovery times in the LMA and ETT groups. We hypothesized that the LMA would be a safe efficient alternative to the ETT.

ELIGIBILITY:
Inclusion Criteria:

* Children 2 to 12 years of age undergoing elective adenotonsillectomy for obstructive sleep apnea or chronic tonsillitis were included in the study.

Exclusion Criteria:

* Exclusion criteria were as follows: Body Mass Index (BMI) greater than 35 and craniofacial anomalies.

Ages: 2 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 131 (Actual)
Dates: Start 2007-12; Primary Completion 2009-08 (Actual); Study Completion 2009-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kelley Dodson, MD, Principal Investigator — Virginia Commonwealth University
Locations (1):
- Virigina Commonwealth University Medical Center, Richmond, Virginia, United States

REFERENCES:
- [Background] Williams PJ, Bailey PM. Comparison of the reinforced laryngeal mask airway and tracheal intubation for adenotonsillectomy. Br J Anaesth. 1993 Jan;70(1):30-3. doi: 10.1093/bja/70.1.30. PMID 8240471

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Endotracheal Tube | Laryngeal Mask Airway
Started | 71 | 60
Completed | 71 | 48
Not Completed | 0 | 12
Not completed — Physician Decision | 0 | 12

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Endotracheal Tube | Laryngeal Mask Airway | Total
Number analyzed (Participants) | 71 | 60 | 131
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 71 | 60 | 131
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 5.5 (2.5) | 5.69 (2.3) | 5.6 (2.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 31 | 25 | 56
  Male | 40 | 35 | 75
Region of Enrollment [Number; unit: participants]
  United States | 71 | 60 | 131

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Laryngospasm
Time Frame: 2 years
Measure: Number; unit: Participants
Arm/Group | Endotracheal Tube | Laryngeal Mask Airway
Number analyzed (Participants) | 71 | 60
Participants | 8 | 6

2. Secondary Outcome: Postanesthesia Recovery Times
Time Frame: After surgery
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Endotracheal Tube | Laryngeal Mask Airway
Number analyzed (Participants) | 71 | 60
minutes | 95.59 (77.72) | 83.50 (58.91)

ADVERSE EVENTS:
Time Frame: No adverse events collected
Description: No adverse events collected.
Arm/Group | Endotracheal Tube | Laryngeal Mask Airway
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No